CLINICAL TRIAL: NCT06920576
Title: Effect of Perioperative Intravenous Infusion of Esketamine or Magnesium Sulphate on Emotional State and Postoperative Pain in Patients Undergoing Nasal Endoscopic Surgery: a Randomised, Controlled Trial
Brief Title: Effects of Esketamine Versus Magnesium Sulfate on Emotional State and Postoperative Pain in Patients Undergoing Nasal Endoscopic Surgery
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Second People's Hospital of Huai'an (Other)
Responsible Party: Principal Investigator, Chenglan Xie, chief physician, The Second People's Hospital of Huai'an
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLXie
Record Dates: First submitted 2025-03-14; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Chronic Rhinosinusitis; Enhanced Recovery After Surgery
Keywords: Esketamine; magnesium sulfate; emotional state; Functional endoscopic sinus surgery
MeSH Terms: interventions — Esketamine; Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization sequence was generated by a computer and handed over in sealed opaque sequentially numbered envelopes. The envelope was opened by anaesthetist not involved in the study and drugs were dispensed as per the allocation card. The configured drugs were then handed over to experienced anaesthetists who were not aware of the subgroups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Esketamine (Experimental): Patients were given intravenous esketamine 0.25 mg/kg 10 min before induction of anaesthesia, followed by continuous pumping at 0.25 mg/(kg-h) until the end of the operation.
  Interventions: Drug: Esketamine
- Magnesium Sulfate (Experimental): Patients in the magnesium sulphate group (Group L) were injected with 30 mg/kg of magnesium sulphate intravenously 10 min before the induction of anaesthesia, followed by continuous pumping at 30 mg/(kg-h) until the end of the operation.
  Interventions: Drug: Magnesium sulfate
- Saline (Placebo Comparator): Control (Group C) patients were pumped with equal volume of saline during the same time period.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Esketamine — Intravenous esketamine 0.25 mg/kg was administered 10 min before induction of anaesthesia, followed by continuous pumping at 0.25 mg/(kg-h) until the end of the operation.
  Arms: Esketamine
Drug: Magnesium sulfate — Intravenous magnesium sulphate 30 mg/kg was administered within 10 min before induction of anaesthesia, followed by continuous pumping at 30 mg/(kg-h) until the end of the operation
  Arms: Magnesium Sulfate
Drug: Saline — Pumping equal volumes of saline over the same time period
  Arms: Saline

SUMMARY:
Functional endoscopic sinus surgery (FESS) is one of the effective modalities for the treatment of Functional endoscopic sinus surgery (FESS) is one of the effective ways to treat chronic sinusitis, which has the advantages of deep approach, light trauma and less pain. However, the operation area involves the nose, eyes and skull.

However, because the operation area involves the nose, eyes and skull, the surrounding tissue structure is complex and rich in blood vessels and nerves, and the use of epinephrine, tissue damage, nerve irritation and other problems during the operation are all related to the treatment of chronic rhinosinusitis.However, because the operation area involves the nose, eyes and skull, the surrounding tissue structure is complex and rich in blood vessels and nerves, and the use of epinephrine, intraoperative tissue damage, nerve stimulation, postoperative inflammation, oedema, bleeding, nasal tamponade can cause stress reactions and The use of adrenaline, intraoperative tissue damage, nerve stimulation, postoperative inflammation, oedema, bleeding, and nasal tamponade can all cause stress reactions and postoperative pain in patients, resulting in anxiety, depression, and sleep disorders, thus reducing the quality of early postoperative recovery and affecting This reduces the quality of early postoperative recovery and affects the rapid recovery of patients. As an NMDA receptor antagonist, esketamine has a strong analgesic effect, fast onset of action and rapid metabolism. As an NMDA receptor antagonist, esketamine has a strong analgesic effect, fast onset of action and fast metabolism, which can effectively alleviate postoperative pain, reduce the need for analgesic drugs, prolong the duration of analgesia, reduce the use of opioids and prevent pain hypersensitivity and preventing nociceptive allergy. In addition, esketamine has been proved to be effective in improving depression and anxiety, as well as sleep disorders. In addition, esketamine has been shown to be effective in improving depression and anxiety and in improving sleep disorders. Based on the action of NMDA receptor antagonists, magnesium sulphate reduces opioid consumption and decreases postoperative pain scores, without increasing opioid use.

Postoperative pain scores, without increasing the risk of opioid side effects, significantly enhancing perioperative analgesia and reducing the need for analgesia 24 hours after surgery. Magnesium sulphate can reduce opioid consumption and postoperative pain scores without increasing the risk of opioid side effects, significantly enhancing perioperative analgesia and reducing the need for analgesia 24 hours after surgery. At present, few studies and experiences have been reported on the use of esketamine and magnesium sulphate in ERAS in otorhinolaryngology, head and neck surgery. At present, there are few studies and experiences on the use of esketamine and magnesium sulfate in ERAS in otolaryngology, head and neck surgery. The aim of this study was to investigate the effects of intravenous infusion of esketamine or magnesium sulfate on postoperative pain and emotional state in patients undergoing nasal endoscopy. The aim of this study was to investigate the effects of intravenous infusion of esketamine or magnesium sulfate on postoperative pain, emotional state and quality of recovery in patients undergoing nasal endoscopy.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of intravenous infusion of esketamine or magnesium sulphate on postoperative pain and quality of recovery in patients undergoing nasal endoscopic surgery.Patients were randomised into group S: intravenous infusion of esketamine (0.25 mg/kg over 10 minutes before induction, then 0.25 mg/kg/h); group L intravenous infusion of magnesium sulphate (30 mg/kg over 10 minutes before induction, then 30 mg/kg/h). The control group was pumped with an equal volume of saline over the same time period. Patients were randomly allocated to the esketamine group, magnesium sulphate group and control group in a 1:1 ratio using a computer generated random sequence and the sealed envelope method. Patients, anaesthetists and researchers observing the results were unaware of the allocation of patients to groups.The patients were routinely fasted for 6 h and abstained from drinking for 2 h preoperatively.The patient was admitted to the room with an open peripheral vein and a continuous infusion of sodium lactate Ringer's solution; cardiac monitoring, pulse rate were routinely performed,oxygen saturation (SpO2) and ECG.A temperature-controlled blanket was used intraoperatively to maintain normothermia. In all three groups, intravenous midazolam 0.05 mg/kg, propofol 1.5 mg/kg, rocuronium bromide 0.6 mg/kg, and sufentanil 0.5 μg/kg were injected.The patients in all three groups were induced with intravenous midazolam 0.05 mg/kg, propofol 1.5 mg/kg, rocuronium bromide 0.6 mg/kg, and sufentanil 0.5 μg/kg for routine fast-channel induction. During anaesthesia maintenance, remifentanil 0.1-0.5 ug/kg/min, sevoflurane (1%-3%) and propofol 4-12 mg/kg were continuously infused in all three groups.Sevoflurane (1%-3%), and Propofol 4-12 mg/kg/h were continuously infused in all three groups. All three groups of patients were connected to a ventilator with 2.0 L/min of pure oxygen for respiratory control, and the parameters were set as follows: tidal volume of 6-8 ml/kg, inspiratory/expiratory ratio of 1:2, and PETCO2 control of 35-40 mmHg. The appropriate depth of anaesthesia was maintained.Maintain appropriate anaesthesia depth (entropy index RE/SE 40～60).At the appropriate depth of anaesthesia, vasoactive drugs (ephedrine, phenylephrine, nitroglycerin) can be administered to regulate blood pressure. Immediately after the procedure, the patient is transferred to the PACU and the endotracheal tube is removed when the patient regains consciousness and can breathe spontaneously. In the PACU, pain severity was measured at fixed intervals on a 10-point numerical rating scale (VAS, 0-10), and postoperative VAS scores >3 were given intravenously with ketorolac aminotriol injection 30 mg for remedial analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists (ASA) classification I-II
* Patients scheduled for FESS under general anaesthesia and with a procedure duration of not less than 30 minutes.

Exclusion Criteria:

* Patients with hypersensitivity to esketamine, magnesium sulphate and other anaesthetic drugs;
* Combined vital organ insufficiency;
* Pregnant and lactating women;
* Those with a history of substance abuse;
* Patients who are unable to understand the study or who are mentally ill;
* Uncontrolled diabetes mellitus, hypertension, hyperthyroidism;
* Failure to understand or cooperate with HADS, SAS, SDS questionnaires, or the Pain Assessment Scale (VAS);
* Those who do not sign the informed consent form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | Preoperative day 1 (PRE1), postoperative day 1 (POD1), postoperative day 3 (POD3)
  The HAD scale consists of 14 items divided into two subscales, anxiety and depression, each subscale contains 7 items, each item is rated on a scale of 0-3, and the total score for anxiety and depression is 0-21.A score of >7 on the HAD scale can be used as a differentiating value for anxiety and/or depression, with scores of 8-10 as mild anxiety and/or depression, 11-14 as moderate anxiety and/or depression, and 15- 21 are classified as severe anxiety and/or depression.
Self-Assessment Scale for Anxiety (SAS) | Preoperative day 1 (PRE1), postoperative day 1 (POD1), postoperative day 3 (POD3)
  The SAS was developed by Zung WW in 1971 to rate patients' subjective feelings of anxiety and changes in treatment.The SAS has 20 items, which are rated on a 4-point scale of 1-4 according to the frequency of symptoms, with 5 reverse scores. The total score was summed to obtain the crude score, and then the crude score was multiplied by 1.25 and the whole number portion was taken to obtain the standard score. The SAS cut-off value was 50 points according to the Chinese normative criteria, with 50-59 points for mild anxiety, 60-69 points for moderate anxiety, and higher than 69 points for severe anxiety.
Depression Self-Rating Scale（SDS） | Preoperative day 1 (PRE1), postoperative day 1 (POD1), postoperative day 3 (POD3)
  The SDS was developed by Zung WW in 1965 to visualise patients' subjective feelings of depression and changes in treatment. The scale is similar to the SAS, with 20 items reflecting an individual's subjective feelings of depression, and is rated on a 4-point scale of 1-4, including 10 reverse scores. The SDS scores were summed to obtain a total crude score, and the standard score was obtained by multiplying the crude score by 1.25 and taking the integer part. The SDS cut-off value according to the Chinese normative scale was 53, with mild depression ranging from 53-62, moderate depression from 63-72, and severe depression above 73.
Pain visual analogue score (VAS) | 2, 24, 48 and 72 hours postoperatively
  The visual analogue scale (VAS) is used for pain assessment. It is widely used in Chinese clinics, and the basic method is to use a 10-cm-long travelling scale with 10 scales on one side and '0' and '10' scores at both ends, with 0 indicating no pain and 10 representing the most severe pain that is difficult to tolerate. 0 is no pain, 1-3 is mild pain; 4-6 is moderate pain, which affects sleep and is still tolerable; 7-10 is severe pain, which is intolerable and affects sleep and appetite.

SECONDARY OUTCOMES:
Intraoperative Propofol and Remifentanil Dosage | intraoperative
  The dosage of propofol and remifentanil was adjusted according to the depth of anesthesia during the operation, and propofol was maintained at a rate of 4~12 mg/kg/h, while remifentanil was maintained at 0.5~1.5 ug/kg/min.
incidence of adverse effects | Postoperative day 1 、Postoperative day 2
  The incidence of perioperative hypotension, hypertension, bradycardia, and tachycardia; PONV; and adverse effects (headache, dizziness, nightmares, sleep disturbances, and mood disorders) was recorded;
Intraoperative phenylephrine, atropine, nitroglycerin, ephedrine dosage | intraoperative
  Vasoactive drugs may be administered at an appropriate depth of anesthesia. When the mean arterial blood pressure(MAP) was >75 mmHg, 20 ug of nitroglycerin was given; when the MAP was less than 60 mmHg, 40 ug of phenylephrine was given preferentially, and 3 mg of ephedrine was given after the ineffective treatment; when the heart rate was less than 45 beats/minute, 0.5 mg of atropine was given.
Heart rate（HR） | Perioperative:entering the operating room, before induction of anesthesia, before intubation, immediately after intubation, start of surgery, end of surgery, at extubation
  perioperative hemodynamic fluctuations
Mean arterial blood pressure(MAP) | Perioperative: entering the operating room, before induction of anesthesia, before intubation, immediately after intubation, start of surgery, end of surgery, at extubation
  perioperative hemodynamic fluctuations

CONTACTS AND LOCATIONS:
Overall Officials: Xie chenglan, PhD, Study Director — The Affiliated Huaian Hospital of Xuzhou Medical University, Huai'an Second Hospital
Locations (1):
- The Affiliated Huaian Hospital of Xuzhou Medical University, Huai'an Second Hospital, Huaian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu H, Hao C, Wang X, Du J, Zhang T, Zhang X. Effect of Intraoperative infusion Magnesium Sulfate Infusion on Postoperative Quality of Recovery in Patients Undergoing Total Knee Arthroplasty: A Prospective, Double-Blind, Randomized Controlled Trial. Drug Des Devel Ther. 2024 Mar 25;18:919-929. doi: 10.2147/DDDT.S444896. eCollection 2024. PMID 38560523
- [Background] Hung KC, Chang LC, Ho CN, Hsu CW, Wu JY, Lin YT, Chen IW. Influence of Intravenous Magnesium Sulfate Infusion on the Subjective Postoperative Quality of Recovery: A Meta-Analysis of Randomized Controlled Trials. Nutrients. 2024 Jul 22;16(14):2375. doi: 10.3390/nu16142375. PMID 39064818
- [Background] Kilic K, Sakat MS, Sahin A, Ahiskalioglu EO, Altunok H. Efficacy of intravenous magnesium sulfate infusion on postoperative pain and quality of recovery for septorhinoplasty: a randomized controlled study. Acta Otolaryngol. 2023 Nov-Dec;143(11-12):979-983. doi: 10.1080/00016489.2023.2289584. Epub 2024 Jan 26. PMID 38108626
- [Background] Zhou Y, Lan X, Wang C, Zhang F, Liu H, Fu L, Li W, Ye Y, Hu Z, Chao Z, Ning Y. Effect of Repeated Intravenous Esketamine on Adolescents With Major Depressive Disorder and Suicidal Ideation: A Randomized Active-Placebo-Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2024 May;63(5):507-518. doi: 10.1016/j.jaac.2023.05.031. Epub 2023 Jul 4. PMID 37414272
- [Background] Yan H, Chen W, Chen Y, Gao H, Fan Y, Feng M, Wang X, Tang H, Yin J, Qian Y, Ding M, Cang J, Miao C, Wang H. Opioid-Free Versus Opioid-Based Anesthesia on Postoperative Pain After Thoracoscopic Surgery: The Use of Intravenous and Epidural Esketamine. Anesth Analg. 2023 Aug 1;137(2):399-408. doi: 10.1213/ANE.0000000000006547. Epub 2023 Jul 14. PMID 37267129
- [Background] Xu Y, He L, Liu S, Zhang C, Ai Y. Intraoperative intravenous low-dose esketamine improves quality of early recovery after laparoscopic radical resection of colorectal cancer: A prospective, randomized controlled trial. PLoS One. 2023 Jun 2;18(6):e0286590. doi: 10.1371/journal.pone.0286590. eCollection 2023. PMID 37267303